CLINICAL TRIAL: NCT00013949
Title: Active Elderly Study
Brief Title: Cardiovascular Vulnerability to Particulate Exposure
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Other Study IDs: 9825-CP-003
Record Dates: First submitted 2001-04-03; First posted 2001-04-04 (Estimated); Last update posted 2006-09-04 (Estimated); Status verified 2006-09

CONDITIONS: Heart Disease; Lung Disease
Keywords: Holter monitoring; ECG; Cardiac; particulate exposure
MeSH Terms: conditions — Heart Diseases; Lung Diseases

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
This project is part of a program project directed toward assessing cardiac effects of particulate and other ambient air pollutants. In this project active elderly adults living in the communities of Boston and Steubenville have attended 12 weekly sessions including approximately 40 minutes of Holter monitoring, blood pressure, and oximetry evaluation before, during, and after outdoor exercise. To investigate the relation of air pollution to cardiac and pulmonary rehabilitation, a second portion of this study involves abstraction of blood pressure and symptom data and downloading of available repeated measures telemetry data in two populations. These populations include: 1) 200 outpatients attending 8 to 36 repeated weekly exercise training sessions in a major hospital cardiac rehabilitation unit.

DETAILED DESCRIPTION:
Approximately 60 subjects have participated fully in Boston and Steubenville in the repeated 40 minute measurement of continuous EKG (Holter), blood pressure, and oximetry. In Steubenville we have also measured exhaled nitrogen oxide, an index of pulmonary inflammation. The exposure monitoring has included outdoor particle mass of PM2.5, outdoor gaseous pollutants, and indoor home and personal monitoring to evaluate the indoor contribution of pollution to health effects.

ELIGIBILITY:
Participants are 50 to 90 years of age, but almost all are 60 and older. They have been enrolled as volunteers from communities in Mission Park, Boston, and Steubenville. Inclusion criteria includes the ability to walk on level ground. Exclusion criteria includes unstable anginal, and baseline EKG patterns such as left bundle branch block that would make difficult the detection of repolarization abnormalities. Participants live at or near the study center which was located in an office or apartment in the apartment building of the majority of the participants.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 1998-09; Study Completion 2004-09

CONTACTS AND LOCATIONS:
Overall Officials: Diane Gold, MD, Study Director — Harvard School of Public Health (HSPH); Frank E Speizer, MD, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States